CLINICAL TRIAL: NCT06857032
Title: Evaluation of the Long-term Safety and Effectiveness of Laser in Situ Keratomileusis (LASIK) in Combination with Corneal UV-riboflavin Crosslinking in Comparison with Classic LASIK for the Correction of Myopia and Myopic Astigmatism
Brief Title: Long-term Safety and Effectiveness of LASIK-Xtra Compared to Conventional LASIK
Acronym: Xtra Lasik
Status: Enrolling by invitation | Type: Observational
Sponsor: University Clinic Frankfurt (Other)
Responsible Party: Principal Investigator, Professor Dr. med. Thomas Kohnen, Professor and Chair, University Clinic Frankfurt
Other Study IDs: 0219-2024
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-09

CONDITIONS: Tomography; Corneal Biomechanics; Manifest Ref; Endothelial Cells; IOP; Optical Coherence Tomography
Keywords: Lasik; Lasik Xtra; Keratectasia; Corneal biomechanics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group 1: Patients treated with Xtralasik

SUMMARY:
Laser in situ keratomileusis (LASIK) is a widely used procedure for the correction of myopia and myopic astigmatism. Despite its high effectiveness and the general safety of the procedure, long-term safety and effectiveness remain a key concern in ophthalmology. A promising further development is the combination of LASIK with corneal UV-riboflavin crosslinking, which promises additional stability of the cornea.1 This study aims to evaluate the long-term safety and effectiveness of this combined method in comparison to classic LASIK. By analysing long-term results, the aim is to gain well-founded insights that will help to optimise the decision on the most suitable procedure for correcting myopia and myopic astigmatism and to ensure the best possible clinical results for patients.

DETAILED DESCRIPTION:
The null hypothesis is that combined laser in situ keratomileusis (LASIK) with corneal UV-riboflavin crosslinking (LASIK-Xtra) has the same long-term safety and effectiveness as classic LASIK for the correction of myopia and myopic astigmatism.

Aim of the study The main objective of this study is to determine whether LASIK-Xtra compared to classic femto-LASIK

1. leads to the same long-term results in terms of postoperative visual acuity,
2. the postoperative spectacle values of both eyes are at least equally stable over several years after the study and
3. the corneal shape and stiffness values do not differ between the procedures after several years.

In addition, possible long-term side effects of the procedures are documented.

The new ophthalmological examination is intended to show that the combination of LASIK-Xtra is at least equally safe and effective compared to the standard variant of Femto-LASIK even after several years.

Safety endpoints:

For the entire study:

1. difference between preoperative and postoperative best corrected visual acuity (BCDVA)
2. occurrence of keratoectatic changes
3. incidence of adverse events

study design

* The retrospective-prospective study includes:

  1. a retrospective collection of examination and surgical results of patients who successfully participated in the study with the clinicaltrials.gov registration number: NCT 03913338 during the study period from 2014 to 2018 at the Department of Ophthalmology of the Goethe University Frankfurt
  2. a prospective follow-up examination in accordance with the standard in ophthalmology to record the visual acuity and eye examination data of patients who were treated between 2014 and 2018 at the Department of Ophthalmology at Goethe University Frankfurt for the correction of myopia and myopic astigmatism in one eye using LASIK-Xtra and in the partner eye using classic femto-LASIK as part of the above-mentioned study
* Performance of non-invasive examinations to assess long-term safety and effectiveness
* De-personalised data collection via MS Excel for Mac (Version 16.53, Microsoft, USA)
* Statistical analysis using SPSS Statistic 29 software (IBM, USA)
* Data security: Data storage is pseudonymised and password-protected

material & methods

Retrospective part:

As part of the study, available visual acuity, results of surgery and examination results already available in the study files of patients who have undergone surgery as part of the NCT 03913338 study will be collected.

No measures will be collected other than those already available in the patient file at the study centre.

Prospective part:

Patients who fulfil the eligibility criteria and agree to participate in the prospective study will be asked to come to the clinic for a single study visit to perform a standard ophthalmological examination in ophthalmology. These include:

Slit lamp examination:

During the study visit, a slit lamp examination will be performed. Particular attention is paid to the cornea. The clarity and quality of the epithelium and stroma will be assessed. All results, including any changes, must be recorded in the patient file and CRF. Photographic documentation is taken.

Subjective refraction:

Basically, subjective refraction is based on the patient's response to changes in lens power and their orientation in relation to the legibility of certain vision charts. This method requires the patient's concentration and co-operation and must be performed by either an optician or ophthalmologist.

Pentacam® AXL Wave (Oculus, Wetzlar, Germany):

This tool is one of the latest ophthalmological measurement devices. The measuring principle is based on a combination of slit illumination and Scheimpflug camera. During data acquisition, the sensors rotate around the eye. It combines the following functions: Scheimpflug tomography, wavefront measurement of the entire eye, objective refraction, axial globe length measurement and retroillumination. All data is collected in one scan within the same measurement axis.

iTrace (Tracey Technologies, Texas, USA): This ray tracing based diagnostic tool offer two different functions: Wavefront measurement and corneal topography. The built-in processor unit allows iTrace (Tracey Technologies, Texas, USA) to calculate additional data (e.g. differentiation between internal optics and total aberration).

Corvis ST® (Oculus, Wetzlar, Germany):

This instrument is a non-contact tonometer that analyses the cornea's response to an air pressure pulse using an ultra-high-speed Scheimpflug camera. The recorded image sequences are used to estimate the intraocular pressure and deformation parameters. All measurements with the Corvis ST are performed in a seated position with the pupil undilated.

Nidek CEM-530 (Nidek Co, Gamagori, Japan):

This is a non-contact spectral microscope for measuring the number and evaluating the shape of the corneal endothelium. Due to the non-contact measurement, there is no risk of corneal infection and no anaesthesia is required.

The measurements are performed by trained and certified staff of the study centre of the Department of Ophthalmology of the Goethe University Hospital.

Patient recruitment:

The patients who successfully participated in the study entitled 'Controlled evaluation of the safety and effectiveness of laser in situ keratomileusis (LASIK) for the correction of myopia and myopic astigmatism in combination with corneal UV riboflavin crosslinking with the KXL system and VibeX Xtra riboflavin eye drops compared to classic LASIK. ' successfully participated in the study period from 2014 to 2018 at the Department of Ophthalmology at Goethe University Frankfurt (clinicaltrials.gov, registration number: NCT 03913338) will be informed about the current study by telephone or electronically via e-mail by employees of the study centre. This involves 19 patients. After giving their consent, they will be invited to the Department of Ophthalmology on an agreed date. This is based on the contact details stored in the study files.

All individuals will be appropriately informed and explicitly informed about the voluntary nature of their participation. Further information can be found in the document 'Patient information and consent form'.

The parameters of the measurements taken during the initial study will be collected from the study file.

6 Data collection The collection of personal patient data is carried out in compliance with the Data Protection Act. The data subject is recorded exclusively via a numerical ID.

statistics The analysis is carried out with SPSS Statistic 29 (IBM, USA). The Shapiro-Wilk test is used to test the normal distribution. The Wilcoxon rank sum test (non-parametric) and the paired t-test (parametric data) are used to determine differences between the different time points. A descriptive data analysis is also carried out.

Case number calculation:

Since the study results are purely descriptive in nature, the sample size is based on the total number of subjects who successfully participated in the study. We expect to collect data from a total of 19 patients (38 eyes) from previous surgeries with LASIK Xtra on one eye and conventional Femto-LASIK on the fellow eye.

Inclusion and exclusion criteria:

Inclusion criteria

For both the retrospective and prospective part of the study:

1. only patients who have successfully participated in the study with the clinicaltrials.gov registration number NCT 03913338 during the study period from 2014 to 2018 at the Department of Ophthalmology of the Goethe University Frankfurt will be included for the study to assess long-term outcomes and safety.
2. adult men or women over the age of 18.
3. subjects must be able to understand the requirements of the study and provide written informed consent.

Exclusion criteria

Applies only to patients participating in the prospective part of the study:

1. employees, relatives or friends of employees of an ophthalmological company or investigational clinic (e.g. investigator, coordinator, technician)

ELIGIBILITY:
Inclusion Criteria:

For both the retrospective and prospective part of the study:

1. only patients who have successfully participated in the study with the clinicaltrials.gov registration number NCT 03913338 during the study period from 2014 to 2018 at the Department of Ophthalmology of the Goethe University Frankfurt will be included for the study to assess long-term outcomes and safety.
2. adult men or women over the age of 18.
3. subjects must be able to understand the requirements of the study and provide written informed consent.

Exclusion Criteria:

Applies only to patients participating in the prospective part of the study:

1. employees, relatives or friends of employees of an ophthalmological company or investigational clinic (e.g. investigator, coordinator, technician)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Xtralasik and participated in the first XtraLasik study
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Manifest refraction | single time point with one and only visit
  Manifest refraction with trial frame

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kohnen, Professor and Doctor, Principal Investigator — University Hospital Frankfurt am Main - Eye clinic
Locations (1):
- University Clinic Frankfurt, Goethe University, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kohnen T, Lwowski C, Hemkeppler E, de'Lorenzo N, Petermann K, Forster R, Herzog M, Bohm M. Comparison of Femto-LASIK With Combined Accelerated Cross-linking to Femto-LASIK in High Myopic Eyes: A Prospective Randomized Trial. Am J Ophthalmol. 2020 Mar;211:42-55. doi: 10.1016/j.ajo.2019.10.024. Epub 2019 Nov 1. PMID 31678559